CLINICAL TRIAL: NCT02916342
Title: Interscalene Brachial Block Versus Combined Supraprascapular: Axillary Nerve Blocks - Respiratory and Acute Pain-related Outcomes
Brief Title: Interscalene Block Versus Combined Supraprascapular: Axillary Nerve Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, PD Dr, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016-00889
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Analgesia; Diaphragm
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interscalene brachial plexus block (Active Comparator): An ultrasound-guided interscalene brachial plexus block will be performed prior to surgery.
  Interventions: Procedure: Interscalene brachial plexus block
- Supraclavicular-axillary nerve blocks (Experimental): A dual supraclavicular-axillary nerve blocks will be performed prior to surgery.
  Interventions: Procedure: Supraclavicular-axillary nerve blocks

INTERVENTIONS:
Procedure: Interscalene brachial plexus block — Patients will receive an ultrasound-guided interscalene brachial plexus block before general anaesthesia.
  Arms: Interscalene brachial plexus block
Procedure: Supraclavicular-axillary nerve blocks — Patients will receive ultrasound-guided supraclavicular and axillary nerve blocks before general anaesthesia.
  Arms: Supraclavicular-axillary nerve blocks

SUMMARY:
The interscalene block provides effective analgesia after shoulder surgery. It consists of injecting local anaesthetic within the brachial plexus, in the interscalene groove, between the anterior and middle scalene muscles. Unfortunately, this technique is associated with respiratory complications such as hemidiaphragmatic paresis due to the spread of the local anaesthetic towards the phrenic nerve that lies close to the brachial plexus, with an incidence up to 100%. The diaphragmatic paresis may be a serious side-effect, especially in patients suffering from a reduced respiratory function such as chronic obstructive pulmonary disease; this entity may even represent a contraindication to the performance of the block.

The shoulder is mainly innervated by the suprascapular and axillary nerves, both of them coming from C5 and C6 branches of the brachial plexus block. Recently, several authors have successfully identified and block these two nerves under ultrasound guidance. Only one randomised controlled trial compared interscalene block with a combination of suprascapular and axillary nerve blocks, and showed inconclusive results probably due to the absence of ultrasound guidance; indeed, analgesia was equivalent at the sixth postoperative hour, while patients with an interscalene block had reduced pain scores in the recovery room. Besides, the authors did not investigate the impact on the respiratory function.

In that randomised controlled trial, the investigators would like to compare the analgesic efficacy and the respiratory outcomes between the interscalene block and the combined suprascapular-axillary nerve blocks.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III;
* 18-85 years of age, inclusive;
* surgery less than 3 hours.

Exclusion Criteria:

* indication for catheter insertion;
* contraindications to brachial plexus block (e.g., allergy to local anaesthetics, malignancy or infection in the area);
* existing neurological deficit in the area to be blocked;
* pregnancy;
* history of neck surgery or radiotherapy;
* severe respiratory disease;
* chest deformity;
* inability to understand the informed consent and demands of the study;
* patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Presence of hemidiaphragmatic paresis (yes/no) | 30 minutes after the injection

SECONDARY OUTCOMES:
Forced expiratory volume in 1 second (liters) | 30 minutes after the injection
Peak expiratory flow (liters/minute) | 30 minutes after the injection
Forced vital capacity (liters) | 30 minutes after the injection
Pain scores in phase 1 recovery (visual analogue scale, 0-10) | 2 hours after surgery
  Visual analogue scale, 0-10
Pain scores at 24 hours postoperatively (visual analogue scale, 0-10) | Postoperative day 1
  Visual analogue scale, 0-10
Intravenous morphine consumption in phase 1 recovery (mg) | 2 hours postoperatively
Oxycodone consumption at 24 hours postoperatively (mg) | Postoperative day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes